CLINICAL TRIAL: NCT06900777
Title: Oral Tacrolimus Capsule Versus Dexamethasone Micro-pulse Therapy for the Treatment of Rapidly Progressing Vitiligo in Children: A Multicenter, Randomized, Controlled Study
Brief Title: Oral Tacrolimus vs Dexamethasone Micro-pulse Therapy in Pediatric Rapidly Progressing Vitiligo: A Multicenter RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJPF-LCY-V202421
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-02

CONDITIONS: Vitiligo; Child; Progressive Disease
Keywords: Tacrolimus; Dexamethasone; Randomized Controlled Trialy; Children; Vitiligo; Safety; Efficacy; Multicenter Study; VASI Score; IGA Score; Immunosuppressive Therapy
MeSH Terms: conditions — Vitiligo; Disease Progression | interventions — Tacrolimus; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized controlled study. Participants are randomly assigned to two groups, receiving tacrolimus or dexamethasone respectively. The study aims to compare the efficacy and safety of the two interventions for treating rapidly progressive vitiligo in children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus Treatment Group (Experimental): Participants in this arm receive oral tacrolimus therapy following the specified dosage and administration schedule in the study protocol for treating rapidly progressive vitiligo in children.
  Interventions: Drug: Tacrolimus
- Dexamethasone Comparison Group (Active Comparator): Participants in this arm receive oral dexamethasone as the comparative intervention, administered according to the study protocol for evaluating its efficacy and safety in treating rapidly progressive vitiligo in children.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Tacrolimus — Participants receive oral tacrolimus capsules at a dosage of 0.1 ± 0.05 mg/kg per day, divided into two administrations. The treatment duration is 24 weeks. Blood drug concentration is monitored to maintain trough levels between 7-15 ng/mL. Safety assessments include regular blood tests (hematology, liver/kidney function, blood glucose) and adverse event tracking.
  Arms: Tacrolimus Treatment Group
Drug: Dexamethasone — Participants receive oral dexamethasone tablets at a dosage of 0.05 ± 0.025 mg/kg per day, administered as a single dose on weekends (Saturday and Sunday). The treatment duration is 24 weeks. Safety evaluations include monitoring of blood parameters (hematology, liver/kidney function, blood glucose), weight, and adrenal function (cortisol, ACTH levels).
  Arms: Dexamethasone Comparison Group

SUMMARY:
This clinical study aims to compare the safety and effectiveness of two treatments-oral Tacrolimus capsules and Dexamethasone micro-pulse therapy-in children aged 4-12 years with rapidly progressing vitiligo. The study is a multicenter, randomized, controlled trial involving 90 participants, who will be divided equally into two groups. One group will receive daily Tacrolimus, while the other will take Dexamethasone on weekends. Over 24 weeks, doctors will monitor improvements in skin repigmentation, side effects, and overall health through regular check-ups and blood tests. The goal is to determine which treatment better controls disease progression and improves quality of life for children with vitiligo.

Key Points:

* For children with rapidly spreading vitiligo.
* Compares two common medications.
* Follows participants for 6 months.
* Focuses on safety and effectiveness.

DETAILED DESCRIPTION:
Background:

Vitiligo is an autoimmune skin condition causing pigment loss, significantly impacting children's well-being. Current treatments like systemic corticosteroids (e.g., Dexamethasone) carry risks of long-term side effects. Tacrolimus, an immunosuppressant with a safer profile in other pediatric conditions, shows promise but lacks evidence for oral use in vitiligo. This trial addresses this gap by comparing Tacrolimus and Dexamethasone.

Study Design:

* Multicenter, randomized, controlled trial across 5 hospitals in China.
* 90 participants (4-12 years) with rapidly progressing non-segmental vitiligo (VIDA score 4).
* Interventions:
* Tacrolimus group: 0.1±0.05 mg/kg/day, divided into two doses.
* Dexamethasone group: 0.05±0.025 mg/kg/weekend pulse dosing.
* Duration: 24 weeks with follow-ups at 4, 8, 12, 16, 20, and 24 weeks.

Outcome Measures:

* Primary: Proportion achieving ≥50% improvement in Vitiligo Area Scoring Index (VASI 50) at 24 weeks.
* Secondary: VASI 75/90 response rates, Investigator Global Assessment (IGA) scores, and safety parameters (blood tests, metabolic panels, adverse events).

Statistical Analysis:

Data will be analyzed using chi-square tests to compare efficacy and safety between groups (significance: p ≤ 0.05). All analyses adhere to intention-to-treat principles.

Ethics & Compliance:

Approved by the Ethics Committee of the First Affiliated Hospital of Air Force Medical University. Informed consent is obtained from all participants' guardians.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-12 years diagnosed with rapidly progressive non-segmental vitiligo (VIDA score ≥4, indicating disease progression within the past 6 weeks).

Total body surface area (BSA) affected by vitiligo between 1% and 50%. Guardians provide written informed consent for the child's participation.

Exclusion Criteria:

* Stable-phase childhood vitiligo. Segmental, mucosal, undetermined, or generalized vitiligo. Systemic immunosuppressive therapy within the past 4 weeks. Known hypersensitivity to tacrolimus, other macrolide drugs, or study drug excipients.

Comorbidities precluding oral tacrolimus use (e.g., severe hepatic/renal dysfunction).

Obesity or systemic diseases (e.g., tuberculosis, acute/chronic infections, hypertension, congenital cardiovascular disease).

Any condition deemed by investigators to increase participant risk or interfere with trial execution.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving VASI 50 Response | 24 weeks
  VASI (Vitiligo Area and Severity Index) 50 response is defined as a 50% or greater reduction in VASI score from baseline. Assessment is conducted by trained dermatologists using standardized VASI scoring criteria.

SECONDARY OUTCOMES:
Change in Vitiligo Area and Severity Index (VASI) Score | 24 weeks
  Calculate the difference between the VASI score at 24 weeks and the baseline VASI score. This reflects the improvement in vitiligo area and severity over the treatment period.
Proportion of Participants Achieving Investigator Global Assessment (IGA) Score Improvement | 24 weeks
  Assess participants' IGA scores at 24 weeks. Participants with an IGA score of "mild" or better (score ≤ 2) are defined as achieving improvement, and the proportion is calculated.
Incidence of Treatment-Emergent Adverse Events | Throughout the 24-week treatment period
  Record all adverse events (e.g., gastrointestinal symptoms, metabolic abnormalities) occurring during the 24-week treatment period. Calculate the incidence rate and analyze their relationship with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Jian, Associate Professor, Principal Investigator — First Affiliated Hospital of Air Force Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided